CLINICAL TRIAL: NCT02653144
Title: Double Blinded Randomized Controlled Study Evaluating the Analgesic Duration of Dexmedetomidine Compared to Dexamethasone as Adjuncts to Single Shot Interscalene Block in Patients Undergoing Ambulatory Shoulder Surgery
Brief Title: the Analgesic Duration of Dexmedetomidine Compared to Dexamethasone as Adjuncts to Single Shot Interscalene Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Amaresh Vydynathan, Assoc. Prof. Anesthesiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-5628
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Opioid Use, Unspecified
Keywords: post operative pain, Dexmedetomidine, Regional anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Anesthetics; Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dexmedetomidine and ropivacaine group (Experimental): In this group, participants will undergo pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation with Ropivacaine 0.5% 20ml + 75mcg of dexmedetomidine
  Interventions: Drug: Ropivacaine; Drug: Dexmedetomidine
- dexamethasone and ropivacaine group (Experimental): In this group, participants will undergo pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation with. Ropivacaine 0.5% 20ml + 4mg dexamethasone
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone
- ropivacaine only group (Active Comparator): In this group, participants will undergo pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation with Ropivacaine 0.5% 20ml (acting as control)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — local anesthetics adjuvants. Ropivacaine 0.5% 20ml. pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation in patients undergoing ambulatory shoulder surgery
  Other Names: anesthetics
Drug: Dexmedetomidine — local anesthetics adjuvants. 75mcg of dexmedetomidine. pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation in patients undergoing ambulatory shoulder surgery
  Other Names: anesthetics
  Arms: dexmedetomidine and ropivacaine group
Drug: Dexamethasone — local anesthetics adjuvants. 4mg dexamethasone. pre-operative single shot interscalene nerve block under ultrasound guidance and peripheral nerve stimulation in patients undergoing ambulatory shoulder surgery
  Other Names: anesthetics
  Arms: dexamethasone and ropivacaine group

SUMMARY:
The purpose of the study is to determine if perineural dexmedetomidine can provide increased prolongation of analgesia when compared to perineural dexamethasone in patients receiving regional block for shoulder surgery. If so, dexmedetomidine may serve as a superior adjunct to peripheral nerve blocks in a rapidly evolving, ambulatory-centered surgical setting.

DETAILED DESCRIPTION:
Currently, the most commonly employed adjunct to peripheral nerve blockade is perineural dexamethasone. In general, at the doses used in regional anesthesia, dexamethasone has a minimal side effect profile. However, while it has been shown to increase duration of analgesia, there have been concerns regarding its neurotoxicity in animal studies. In addition, dexamethasone has the potential to cause hyperglycemia in patients with impaired glucose metabolism as well as perineal pain and pruritis when administered peripherally.

Dexmedetomidine is a highly selective alpha-2 agonist that is commonly used in patients undergoing anesthesia or requiring sedation in a non-operative setting. As a peripherally administered medication, it has both sedating and analgesic properties, as well as the added benefit of avoidance of respiratory depression. Although it can rarely produce cardiac depression at high doses, its side effect profile is otherwise minimal and is generally very well tolerated by most patients. When administered peripherally, dexmedetomidine has most commonly been associated with side effects such as hypotension, respiratory depression, and bradycardia - although all at significantly higher doses than planned in our study. The safe use of perineural dexmedetomidine together with local anesthetics has been described on numerous occasions. Nevertheless, although it has been shown to potentiate peripheral nerve blockade and prolong duration of analgesia in various studies , it remains rarely used as an adjunct to regional anesthesia.

ELIGIBILITY:
Inclusion Criteria :

* ASA 1 and 2
* 18-60 years old
* Patients scheduled for ambulatory arthroscopic or open surgery

Exclusion Criteria:

* ASA 3 and 4
* Pre-existing pain disorder
* Regular consumption of chronic pain medication
* Anatomical abnormalities of upper extremity
* Known allergy or hypersensitivity to Ropivacaine or other amide local anesthetics
* Known allergy to dexmedetomidine
* Coagulopathy
* Uncontrolled Diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amaresh Vydyanathan, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Background] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360
- [Background] Fritsch G, Danninger T, Allerberger K, Tsodikov A, Felder TK, Kapeller M, Gerner P, Brummett CM. Dexmedetomidine added to ropivacaine extends the duration of interscalene brachial plexus blocks for elective shoulder surgery when compared with ropivacaine alone: a single-center, prospective, triple-blind, randomized controlled trial. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):37-47. doi: 10.1097/AAP.0000000000000033. PMID 24317234
- [Background] Esmaoglu A, Yegenoglu F, Akin A, Turk CY. Dexmedetomidine added to levobupivacaine prolongs axillary brachial plexus block. Anesth Analg. 2010 Dec;111(6):1548-51. doi: 10.1213/ANE.0b013e3181fa3095. Epub 2010 Oct 1. PMID 20889939
- [Background] Ironfield CM, Barrington MJ, Kluger R, Sites B. Are patients satisfied after peripheral nerve blockade? Results from an International Registry of Regional Anesthesia. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):48-55. doi: 10.1097/AAP.0000000000000038. PMID 24310051
- [Background] Rasmussen SB, Saied NN, Bowens C Jr, Mercaldo ND, Schildcrout JS, Malchow RJ. Duration of upper and lower extremity peripheral nerve blockade is prolonged with dexamethasone when added to ropivacaine: a retrospective database analysis. Pain Med. 2013 Aug;14(8):1239-47. doi: 10.1111/pme.12150. Epub 2013 Jun 11. PMID 23755801
- [Background] Williams BA, Schott NJ, Mangione MP, Ibinson JW. Perineural dexamethasone and multimodal perineural analgesia: how much is too much? Anesth Analg. 2014 May;118(5):912-4. doi: 10.1213/ANE.0000000000000203. No abstract available. PMID 24781562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
Started | 30 | 28 | 31
Completed | 30 | 28 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group | Total
Number analyzed (Participants) | 30 | 28 | 31 | 89
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54 [49 to 59] | 52 [45 to 57] | 52 [39 to 57] | 53.5 [45 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 12 | 44
  Male | 12 | 14 | 19 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Inter-Quartile Range); unit: kg/m2] | 31 [27 to 33] | 29 [26.2 to 31.2] | 29 [25 to 32] | 29 [26 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirements (Morphine Equivalents)
Description: How much opioid did patient ask for within 24 hours post op
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: morphine milligram equivalent
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
Number analyzed (Participants) | 30 | 28 | 31
morphine milligram equivalent | 15 [0 to 30] | 15 [0 to 20.6] | 22.5 [10 to 30]

2. Secondary Outcome: Opioid Requirements (Morphine Equivalents)
Description: How much opioid did patient ask for within 48 hours post op
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: morphine milligram equivalent
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
Number analyzed (Participants) | 30 | 28 | 31
morphine milligram equivalent | 52.5 [30 to 75] | 30 [22 to 50.6] | 40 [25 to 67.5]

3. Secondary Outcome: Time to Discharge From PACU to First Opioid Consumption
Description: How long after surgery does patient take to ask for opioid to manage pain
Time Frame: 24-48 hours after surgery
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
Number analyzed (Participants) | 30 | 28 | 31
minutes | 1280 [977 to 1434] | 1130 [854 to 1325] | 900 [609 to 1348]

4. Secondary Outcome: Return of Motor and Sensory Function
Description: Between 24 to 48 hours after surgery, questionnaire will be used to determine if motor and sensory function have returned.
Time Frame: 24-48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
Number analyzed (Participants) | 30 | 28 | 31
minutes | 1280 [977 to 1434] | 1130 [854 to 1325] | 900 [609 to 1348]

ADVERSE EVENTS:
Time Frame: Subjects were followed up to 48 hours after operations
Arm/Group | Dexmedetomidine and Ropivacaine Group | Dexamethasone and Ropivacaine Group | Ropivacaine Only Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02653144/Prot_SAP_000.pdf